CLINICAL TRIAL: NCT04355312
Title: Using INDOcyanine Green to Analyse Ovarian Vascularization After Ovarian Laparoscopic CYStectomy
Acronym: KYSINDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre Imagerie Cellulaire Santé, Faculté Médecine et Pharmacie, CLERMONT FERRAND (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI 2019 GREMEAU; 2019-001966-14 (Other: 2019-001966-14)
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Ovarian Cysts; Endometriosis; Fertility
Keywords: Laparoscopic Ovarian Cystectomy; Indocyanine Green to study ovarian vascularization; Fertility
MeSH Terms: conditions — Ovarian Cysts; Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kysindo (Experimental): Group of 45 patients with short-term desire for pregnancy who will undergo laparoscopic ovarian cystectomy with use of indocyanine green. Evaluation of the ovarian reserve preoperatively and longitudinal cohort follow-up after surgery at 6 months and 12 months. Analysis by a new imaging technique.
  Interventions: Diagnostic Test: Use of Indocyanine Green in laparoscopic ovarian cystectomy

INTERVENTIONS:
Diagnostic Test: Use of Indocyanine Green in laparoscopic ovarian cystectomy — During intraperitoneal cystectomy or Plasmajet destruction of the cyst, as a benign organic cyst requiring surgical treatment, peroperatively, at the end of the cystectomy procedure, injection by the anesthetist on a peripheral venous route of a bolus of Indocyanine green diluted 0.2mg / kg. Installation of the SPIES camera system (KARL STORZ GmbH & Co.KG, Tuttlingen, Germany).
  Evaluation of the degree of fluorescence at the location of cystectomy or destruction of the cyst.
  A fluorescence score between 0 and 4 (on the model of a Likert scale) will be used for the evaluation of fluorescence.
  A second reading of the Likert scale results will be carried out by a second inspector so that the score is as objective as possible. Then, second evaluation technique realized by the METAMORPH software, which will assign a raw and objective score according to the fluorescence visualized.

SUMMARY:
To evaluate the feasibility of using Indocyanine Green in the laparoscopic surgical treatment of benign organic ovarian cysts (dermoid, serous, mucinous and endometriotic) in patients with a short-term desire for pregnancy. The use of Indocyanine Green during this surgery could allow early evaluation of the absence of alteration of the underlying ovary by the cystectomy. To do so, the fluorescence scores (indocyanine green staining) need to be compared to the ovarian reserve of the patient, previously verified intraoperatively and postoperatively at M6 and M12, these scores being determined according to the vascularization visualized in laparoscopy and established both by a double visual notation (Likert scale) and by a computer software (METAMORPH) objective notation. This procedure would, in patients with fertility disorders or wishing for pregnancy in the short run, reassure them about their reproductive potential immediately after the intervention. In the event of poor staining, if correlated by a decrease in ovarian reserve, the concerned patients could be referred to a MPA treatment facility much earlier in the postoperative period or, if no desire for immediate pregnancy, towards fertility preservation methods.

DETAILED DESCRIPTION:
The study will be open to any patient meeting the inclusion / exclusion criteria, scheduled for intraperitoneal cystectomy or cyst destruction using Plasmajet, corresponding to a benign organic cyst requiring surgical treatment according to current recommendations.

It will proceed as follows:

* Recruitment of patients during the preoperative consultation. The information form will be given to the patient.
* The day before the intervention: Inclusion proposed to the patient after re-explanation of the objectives and the progress of the study, submission of the consent form for the patient to sign. Realization of an ultrasound with count of antral follicles, and description of the ovarian cyst (size, aspect, IOTA criteria). Performing a blood test with AMH measurement to assess the preoperative ovarian reserve.
* The day of the intervention: Intraoperative, injection at the end of the procedure of a bolus of indocyanine green intravenously. Studied through an infrared camera system - the SPIES system (KARL STORZ GmbH & Co. KG, Tuttlingen, Germany) - fluorescence within the ovary will bring out the vascularization of the area of cystectomy or destruction of the cyst. Evaluation of the degree of fluorescence (between 0 and 4, on the model of a Likert scale) carried out at the area of cystectomy or destruction of the cyst. Then, the second evaluation technique using the METAMORPH software will assign a raw and objective score according to the fluorescence visualized. The 2 evaluation results will be compared with each other.
* Postoperatively: there will be no special clinical or biological monitoring. If undesirable effects related to Indocyanine Green occur, they will be noted.
* After discharge, as part of her standard follow-up for short-term desire for pregnancy: she will have a postoperative consultation planned 1 month after the intervention, followed by examination at 6 months and 12 months with an ultrasound for evaluation CFA and blood work with AMH.

Any natural pregnancy will be noted.

ELIGIBILITY:
Inclusion Criteria:

* An adult woman of childbearing potential who has a desire for short-term pregnancy, under the age of 42, to undergo laparoscopic accessible surgical treatment (<10 cm) for a benign organic ovarian cyst (serous, mucinous, dermoid or endometriotic) whose diagnosis was made on imaging (ultrasound or MRI).
* Patient able to provide informed consent to her participation in the study.
* Patient covered by the " Sécurité Social " insurance system.

Exclusion Criteria:

* Adult patient under protection, tutorship or curatorship.
* Refusal of the patient or poor understanding of the French language.
* Known allergy to iodine.
* Current pregnancy or breastfeeding

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Fluorescence uptake or not at the area of cystectomy (binary criterion) | Inoperative
  A fluorescence score based on a Likert scale will be used. The presence of fluorescence will correspond to a success, defined by a value on the scale strictly greater than 0. The absence of fluorescence will be a failure, defined as equal to 0. The judgment criterion will therefore be binary (fluorescence uptake or no at the area of cystectomy), allowing the feasibility judgement.

SECONDARY OUTCOMES:
METAMORPH Score | In immediate postoperative
  Automatic and objective allocation by the METAMORPH software of a raw score according to the fluorescence visualized.
Rate of Side Effects | In per and immediate postoperative
  Accounting for side effects and the occurrence of post-operative complications related to the injection of Indocyanine green.
Added time | Immediate post operativ
  Estimation of the protocol-related time added to the total operating time.
AMH dosage | Preoperatively
  Evaluation of the ovarian reserve biological by AMH dosage in comparison of the fluorescence scores. Study of natural fertility in the year following the cystectomy in the patients wishing for pregnancy.
AMH dosage | Month 6
  Evaluation of the ovarian reserve biological by AMH dosage in comparison of the fluorescence scores. Study of natural fertility in the year following the cystectomy in the patients wishing for pregnancy.
AMH dosage | Month 12
  Evaluation of the ovarian reserve biological by AMH dosage in comparison of the fluorescence scores. Study of natural fertility in the year following the cystectomy in the patients wishing for pregnancy.
Evaluation of the ovarian reserve by ultrasound by CFA | Preoperatively
  Evaluation of the ovarian reserve biological by by ultrasound by CFA in comparison of the fluorescence scores. Study of natural fertility in the year following the cystectomy in the patients wishing for pregnancy.
Evaluation of the ovarian reserve by ultrasound by CFA | Month 6
  Evaluation of the ovarian reserve biological by by ultrasound by CFA in comparison of the fluorescence scores. Study of natural fertility in the year following the cystectomy in the patients wishing for pregnancy.
Evaluation of the ovarian reserve by ultrasound by CFA | Month 12
  Evaluation of the ovarian reserve biological by by ultrasound by CFA in comparison of the fluorescence scores. Study of natural fertility in the year following the cystectomy in the patients wishing for pregnancy.
Number of Participants with Pregnancy | Month 6
  Study of natural fertility in the year following the cystectomy in the patients wishing for pregnancy.
Number of Participants with Pregnancy | Month 12
  Study of natural fertility in the year following the cystectomy in the patients wishing for pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie GREMEAU, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France